CLINICAL TRIAL: NCT02662452
Title: Randomized, Double-blind, Placebo-controlled, First-in-Human Study of GLPG2222 in Healthy Male Subjects
Brief Title: First-in-Human Single and Multiple Dose of GLPG2222
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GLPG2222-CL-101; 2015-004466-29 (EudraCT Number)
Record Dates: First submitted 2016-01-20; First posted 2016-01-25 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-01

CONDITIONS: Healthy
MeSH Terms: interventions — GLPG2222

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- GLPG2222 single dose (Experimental): Single dose of GLPG2222 oral suspension
  Interventions: Drug: GLPG2222 single dose
- Placebo single dose (Placebo Comparator): Single dose of placebo oral suspension
  Interventions: Drug: Placebo single dose
- GLPG2222 multiple doses (Experimental): Multiple doses of GLPG2222 oral suspension
  Interventions: Drug: GLPG2222 multiple doses
- Placebo multiple doses (Placebo Comparator): Multiple doses of placebo oral suspension
  Interventions: Drug: Placebo multiple doses

INTERVENTIONS:
Drug: GLPG2222 single dose — single ascending doses, oral suspension
  Arms: GLPG2222 single dose
Drug: Placebo single dose — single doses, oral suspension, matching placebo
  Arms: Placebo single dose
Drug: GLPG2222 multiple doses — multiple ascending doses, daily for 14 days, oral suspension
  Arms: GLPG2222 multiple doses
Drug: Placebo multiple doses — multiple doses, daily for 14 days, oral suspension, matching placebo
  Arms: Placebo multiple doses

SUMMARY:
The purpose of this First-in-Human study is to evaluate the safety and tolerability after single ascending oral doses of GLPG2222 given to healthy subjects, compared to placebo (Part 1). Also, the safety and tolerability of multiple ascending oral doses of GLPG2222 given to healthy subjects daily for 14 days compared to placebo, will be evaluated (Part 2).

Furthermore, during the course of the study after single and multiple oral dose administrations, the amount of GLPG2222 present in the blood and urine (pharmacokinetics) will be characterized.

The potential of cytochrome P450 (CYP)3A4 interaction after repeated dosing with GLPG2222 will be explored as well.

ELIGIBILITY:
Inclusion Criteria:

* Males between 18-50 years of age
* Subjects must have a body mass index between 18-30 kg/m²
* Subjects must be judged to be in good health based upon the results of a medical history, physical examination, vital signs, 12-lead electrocardiogram and laboratory profile
* Subjects must have a screening spirometry with forced expiratory volume in 1 second ≥80% of predicted values for age, gender and height (Part 1 only)

Exclusion Criteria:

* A subject with a known hypersensitivity to study drug ingredients or a significant allergic reaction to any drug
* Concurrent participation or participation within 8 weeks prior to the initial study drug administration in a drug/device or biologic investigational research study
* A subject with active drug or alcohol abuse within 2 years prior to the initial study drug administration
* Current sexually active (and/or child wish) male; a contraception method must be used

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2016-01; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change versus placebo in number of subjects with adverse events | Between screening and 7-10 days after the last dose
  To evaluate the safety and tolerability of GLPG2222 in comparison with placebo after a single oral dose and multiple oral doses in healthy subjects in terms of adverse events
Change versus placebo in number of subjects with abnormal laboratory parameters | Between screening and 7-10 days after the last dose
  To evaluate the safety and tolerability of GLPG2222 in comparison with placebo after a single oral dose and multiple oral doses in healthy subjects in terms of abnormal laboratory parameters
Change versus placebo in number of subjects with abnormal vital signs | Between screening and 7-10 days after the last dose
  To evaluate the safety and tolerability of GLPG2222 in comparison with placebo after a single oral dose and multiple oral doses in healthy subjects in terms of abnormal vital signs
Change versus placebo in number of subjects with abnormal electrocardiogram | Between screening and 7-10 days after the last dose
  To evaluate the safety and tolerability of GLPG2222 in comparison with placebo after a single oral dose and multiple oral doses in healthy subjects in terms of abnormal electrocardiogram
Change versus placebo in number of subjects with abnormal physical examination | Between screening and 7-10 days after the last dose
  To evaluate the safety and tolerability of GLPG2222 in comparison with placebo after a single oral dose and multiple oral doses in healthy subjects in terms of abnormal physical examination
Change versus placebo in number of subjects with abnormal pulmonary function | Between screening and 4 days after the last dose (Part 1 only)
  To evaluate the safety and tolerability of GLPG2222 in comparison with placebo after a single oral dose and multiple oral doses in healthy subjects in terms of abnormal pulmonary function as measured by spirometry

SECONDARY OUTCOMES:
The amount of GLPG2222 in plasma | Between Day 1 predose and 48 hours after the (last) dose
  To characterize the amount of GLPG2222 in plasma over time - pharmacokinetics (PK) - after a single oral dose and multiple oral doses in healthy subjects
The amount of GLPG2222 in urine | Between Day 1 predose and 24 hours after the (last) dose
  To characterize the amount of GLPG2222 in urine over time - pharmacokinetics (PK) - after a single oral dose and multiple oral doses in healthy subjects
Ratio of 6-b-hydroxycortisol/cortisol in urine | Twelve hours before dosing on Day 1 and Day 14
  To assess the potential of CYP3A4 interaction after repeated oral dosing with GLPG2222 by means of the ratio of 6-b-hydroxycortisol/cortisol in urine

CONTACTS AND LOCATIONS:
Overall Officials: Kirsteen Donaldson, MD, Study Director — Galapagos NV
Locations (1):
- SGS LSS Clinical Pharmacology Unit Antwerp, Antwerp, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No